CLINICAL TRIAL: NCT04676334
Title: CATCH-R: A Rollover Study to Provide Continued Access to Clinical Therapy With Rucaparib
Brief Title: CATCH-R: A Rollover Study to Provide Continued Access to Rucaparib
Acronym: CATCH-R
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: pharmaand GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-111; 2020-001538-37 (EudraCT Number)
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer; Ovarian Cancer; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Other Solid Tumor
Keywords: rucaparib; mCRPC; ovarian cancer; PARP inhibitor; PARPi; CRPC; solid tumor; Clovis Oncology; Antineoplastic agents; Genital Neoplasms, male; Prostatic Neoplasms; Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Genital Neoplasms, Male; Prostatic Neoplasms | interventions — rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rucaparib (Experimental): Rucaparib administered at dose and schedule last taken in parent study, or per investigator decision.
  Interventions: Drug: Rucaparib
- Long-term Follow-up (No Intervention): Participants discontinued rucaparib treatment and were in long-term follow-up in the parent study.

INTERVENTIONS:
Drug: Rucaparib — Rucaparib will be administered daily.
  Other Names: CO-338; Rubraca
  Arms: Rucaparib

SUMMARY:
This protocol is designed to provide participants currently benefiting from rucaparib treatment in a Clovis-sponsored clinical study with continued access to treatment for as long as they continue to benefit. Participants in long-term follow-up (LTFU) in a parent study may also enroll in this study for continued data collection, as applicable based on parent study objectives.

DETAILED DESCRIPTION:
Participants enrolled in this study are required to have completed an End-of-Treatment (EOT) Visit with associated assessments as specified in the Clovis-sponsored parent study (NCT01891344; NCT01968213; NCT02855944). Participants who are no longer receiving treatment and are in LTFU in the parent study (NCT02855944) may enroll into the LTFU portion of this study, as applicable based on parent study objectives, without repeating the EOT visit.

The starting dose of rucaparib administered at initiation of this study will be the same as the last dose received in the parent study, or as deemed appropriate by the investigator and based on available dose strength tablets. The first treatment in the rollover study will begin at the next scheduled treatment visit following the EOT Visit in the parent study.

Participants enrolled to receive continued rucaparib may be treated until disease progression, as assessed by the investigator, unacceptable toxicity, withdrawal of consent, death, loss to follow-up, or study closure by the sponsor. If a participant demonstrates disease progression per investigator assessment while receiving treatment with rucaparib but continues to derive clinical benefit, then continuation of treatment beyond progression is permitted based on investigator decision and participant consent. If a participant continues treatment post-progression, all study assessments should be continued per institutional standard of care. The participant should be discontinued from treatment once it is clear that no further clinical benefit can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a Clovis-sponsored study of rucaparib that is being closed
* Either: (a) Is currently tolerating a rucaparib treatment regimen in the parent study with evidence of clinical benefit, as assessed by the investigator, or (b) Has discontinued treatment and is being followed for collection of LTFU data in the parent study
* Demonstrated compliance with the parent study requirements, as assessed by the investigator, and participant is able and willing to comply with the necessary study visits and assessments as part of the rollover study
* Provided written informed consent prior to enrolling in this rollover study

Exclusion Criteria (applicable only to participants considered for continuation of rucaparib treatment):

* Participant has been permanently discontinued from study treatment in the parent study for any reason
* Pregnant or breastfeeding female patients
* Presence of any other condition that may, in the opinion of the investigator, make the participant inappropriate for continuation of rucaparib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- Canada (5):
  - London Regional Cancer Centre, London, Ontario
  - Institut De Recherche De L'Hospital D'Ottawa, Ottawa, Ontario
  - Princess Margaret Hospital - Toronto, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
- Israel (2):
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
- Italy (5):
  - Istituto per la Ricerca e la Cura del Cancro Istituto di Candiolo, Candiolo, Torino
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale per lo studio e la cura dei tumori "Fondazione Pascale" Oncologia Medica, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Poland (2):
  - Białostockie Centrum Onkologii im. Marii Skłodowskiej-Curie, Bialystok, Podlaskie Voivodeship
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
- Russia (9):
  - Republic Clinical Oncology Dispensary of the Ministry of Healthcare of Republic of Bashkortostan, Ufa, Bashkortosta
  - State Healthcare Institution Oncologic Dispensary No. 2 - Health Department of Krasnodar Region, Sochi, Krasnodarskiy Kray
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangel'sk, Primorskiy (Maritime) Kray
  - Republican oncological dispensary of Republic of Mordovia, Saransk, Respublika Mordoviya
  - Pyatigorsk Oncological Dispensary, Pyatigorsk, Stavropol Kray
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Omsk Regional Clinical Oncologic Dispensary, Omsk
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Almazov National Medical Research Centre, Saint Petersburg
- United Kingdom (2):
  - University College London Hospitals, London, England
  - East and North Hertfordshire NHS Trust, Middlesex, England

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only serious adverse event (SAE) and adverse event of special interest (AESI) safety data were collected, other (non-serious) adverse events (AEs) were not collected. Safety data were collected only for the Rucaparib arm (participants who received rucaparib during this study); safety data were not collected for the Long-term Follow-up arm (participants who did not receive rucaparib during this study).
Groups:
- Rucaparib: Participants received rucaparib at a dose and schedule last taken in the parent study, or per investigator decision.
Period: Overall Study
Arm/Group | Rucaparib | Long-term Follow-up
Started | 20 | 14
Received at Least 1 Dose of Study Drug | 20 | 0
Completed | 20 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Population: all participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rucaparib | Long-term Follow-up | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.92) | 60.5 (7.04) | 59.7 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 17 | 9 | 26
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 12 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing SAEs and AESIs
Description: An SAE was any untoward medical occurrence that occurred at any dose, or after informed consent was given and prior to dosing if the SAE was related to a study procedure, that: resulted in death; was life-threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly or birth defect; or was an important medical event that may not have resulted in death, was not life-threatening, or did not require hospitalization but may be considered an SAE, based on appropriate medical judgment. An AESI was defined as any AE of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate. A summary of all SAEs regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: From first dose of rucaparib through 28 days after receiving last dose of rucaparib (approximately 20 months)
Population: Safety Population: all participants who received rucaparib during the study (Rucaparib arm), safety data were not collected for the Long-term Follow-up arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Rucaparib
Number analyzed (Participants) | 20
Participants
  SAEs | 2
  AESIs | 0

ADVERSE EVENTS:
Time Frame: From first dose of rucaparib through 28 days after receiving last dose of rucaparib (approximately 20 months)
Description: Only SAE and AESI safety data were collected, other (non-serious) AEs were not collected. Safety data were collected only for the Rucaparib arm (participants who received rucaparib during this study); safety data were not collected for the Long-term Follow-up arm (participants who did not receive rucaparib during this study). Data reported for Safety Population: all participants who received rucaparib during the study.
Arm/Group | Rucaparib
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rucaparib (N=20)
Fatigue (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
Only SAE and AESI safety data were collected, other (non-serious) AEs were not collected. Safety data were collected only for the Rucaparib arm (participants who received rucaparib during this study); safety data were not collected for the Long-term Follow-up arm (participants who did not receive rucaparib during this study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (1):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT04676334/Prot_001.pdf